CLINICAL TRIAL: NCT01938937
Title: The Effect of Acute Transcranial Bright Light on Anxiety Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Valkee Oy (Industry)
Responsible Party: Principal Investigator, Heidi Jurvelin, PhD student, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANX-a
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Transcranial bright light exposure (Experimental): Transcranially administered bright light exposure for 12 minutes
  Interventions: Device: Transcranial bright light device
- Transcranial sham exposure (Sham Comparator): Transcranially administered sham exposure for 12 minutes
  Interventions: Device: Transcranial sham device

INTERVENTIONS:
Device: Transcranial bright light device
  Other Names: Valkee npt 1100
  Arms: Transcranial bright light exposure
Device: Transcranial sham device
  Other Names: Valkee npt 1100
  Arms: Transcranial sham exposure

SUMMARY:
The purpose of this study is to determine if transcranially administered bright light has acute effect on anxiety symptoms.

DETAILED DESCRIPTION:
Subjects (n=30) with anxiety symptoms will be recruited into the study. To be included into the study, subjects have to get at least seven points in BAI(Becks Anxiety Inventory). At the beginning of the study subject will be randomly assigned to 12 minutes of acute transcranial bright light or placebo exposure group. Anxiety symptoms will be measured using Spielberger State-Trait Anxiety Inventory (STAI, form Y1)self-rating questionnaire just before and 10 and 110 minutes after the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Subject can read and understand the study protocol
* The written informed consent is obtained from subject
* Subject's BAI total score >= 7

Exclusion Criteria:

* Subject has a lifetime psychotic disorder
* Subject abuses substance or has a dependence
* Subject has had suicidal idealization during the past month
* Subject use psychotropic medications
* Subject has unstable somatic disease
* Subject has used bright-light therapy for the current episode
* Subject is pregnant
* Subject is a relative of a member of research team
* Subject has used transcranial light treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in total score of STAI-Y1 | just before exposure, 10 minutes and 110 minutes after the exposure
  STAI-Y1 (Spielberger State-Trait Anxiety Inventory, form Y1)

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University, Oulu, Finland